CLINICAL TRIAL: NCT03368859
Title: Phase 2 Study Comparing Efficacy and Safety of ABT-165 Plus FOLFIRI vs Bevacizumab Plus FOLFIRI in Metastatic Colorectal Cancer Previously Treated With Fluoropyrimidine, Oxaliplatin and Bevacizumab
Brief Title: A Study of ABT-165 Plus FOLFIRI vs Bevacizumab Plus FOLFIRI in Subjects With Metastatic Colorectal Cancer Previously Treated With Fluoropyrimidine, Oxaliplatin and Bevacizumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study may continue
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-064; 2017-003669-87 (EudraCT Number)
Record Dates: First submitted 2017-12-06; First posted 2017-12-11 (Actual); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Cancer
Keywords: cancer; colorectal cancer; ABT-165; FOLFIRI; Bevacizumab; bowel cancer; metastatic colorectal cancer; metastatic colorectal
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms | interventions — Leucovorin; Fluorouracil; Bevacizumab; ABT-165; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABT-165 plus FOLFIRI (Experimental): ABT-165 plus FOLFIRI (irinotecan, leucovorin, fluorouracil).
  Interventions: Drug: Leucovorin; Drug: Fluorouracil - bolus; Drug: Fluorouracil - infusion; Drug: ABT-165; Drug: Irinotecan
- Bevacizumab plus FOLFIRI (Active Comparator): Bevacizumab plus FOLFIRI (irinotecan, leucovorin, fluorouracil).
  Interventions: Drug: Leucovorin; Drug: Fluorouracil - bolus; Drug: Bevacizumab; Drug: Fluorouracil - infusion; Drug: Irinotecan

INTERVENTIONS:
Drug: Leucovorin — Intravenous
  Other Names: Folinic Acid
Drug: Fluorouracil - bolus — Intravenous
  Other Names: 5-FU
Drug: Bevacizumab — Intravenous
  Other Names: Avastin
  Arms: Bevacizumab plus FOLFIRI
Drug: Fluorouracil - infusion — Intravenous
  Other Names: 5-FU
Drug: ABT-165 — Intravenous
  Arms: ABT-165 plus FOLFIRI
Drug: Irinotecan — Intravenous
  Other Names: Irinotecan hydrochloride

SUMMARY:
A study to evaluate the efficacy and tolerability of ABT-165 plus FOLFIRI compared to bevacizumab plus FOLFIRI in participants with previously treated metastatic adenocarcinoma of the colon or rectum.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically confirmed metastatic adenocarcinoma of the colon or rectum.

  * Primary tumor has been resected > 3 months prior to randomization.
* At least 1 lesion on a computed tomography (CT) scan (preferred) or magnetic resonance imaging (MRI) that is measurable as defined by Response Evaluation Criteria In Solid Tumors (RECIST), Version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance score of 0 or 1.
* Progression following treatment with fluoropyrimidine/oxaliplatin/bevacizumab-regimen in the metastatic setting.
* Adequate hematologic, renal and hepatic function.

Exclusion Criteria:

* Any prior therapy with irinotecan
* Unresolved clinically significant toxicities from prior anticancer therapy, defined as any Common Terminology Criteria for Adverse Events (CTCAE) => Grade 2
* Clinically significant conditions that increase the risk for antiangiogenic therapy.
* History of any of the following during first-line therapy with a bevacizumab-containing regimen: arterial thrombotic/thromboembolic event, bowel perforation, Grade 4 hypertension, Grade 3 proteinuria or Grade 3 - 4 bleeding event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (65):
- United States (46):
  - Ironwood Cancer & Res Ctr /ID# 200044, Chandler, Arizona
  - Highlands Oncology Group /ID# 169289, Fayetteville, Arkansas
  - City of Hope /ID# 200501, Duarte, California
  - St. Joseph Heritage Healthcare /ID# 200100, Fullerton, California
  - USC Norris Cancer Center /ID# 200410, Los Angeles, California
  - Hoag Memorial Hosp Presbyterian /ID# 202661, Newport Beach, California
  - Torrance Health Association (DBA)Torrance Memorial Physician Network/Cancer Care /ID# 202488, Redondo Beach, California
  - UC Davis Comprehensive Cancer Center - Main /ID# 207227, Sacramento, California
  - Pacific Central Coast Health Centers-SLO Oncology and Hematology Health Center /ID# 201215, San Luis Obispo, California
  - Central Coast Medical Oncology /ID# 200227, Santa Maria, California
  - University of California, Los /ID# 169294, Santa Monica, California
  - Kaiser Permanente, Waterpark III Institute for Health Research /ID# 200801, Aurora, Colorado
  - Georgetown University Hospital /ID# 202903, Washington D.C., District of Columbia
  - Florida Cancer Specialist - South /ID# 203796, Fort Myers, Florida
  - Florida Cancer Specialists-Panhandle /ID# 203787, Tallahassee, Florida
  - IACT Health /ID# 169292, Columbus, Georgia
  - Ingalls Memorial Hosp /ID# 169892, Harvey, Illinois
  - Illinois Cancer Care, PC /ID# 202189, Peoria, Illinois
  - Fort Wayne Medical Oncology /ID# 201616, Fort Wayne, Indiana
  - Cancer Center of Kansas /ID# 200627, Wichita, Kansas
  - Norton Cancer Institute /ID# 200674, Louisville, Kentucky
  - Ochsner Clinic Foundation-New Orleans /ID# 169291, New Orleans, Louisiana
  - Whiteside Institute for Clinic /ID# 200802, Duluth, Minnesota
  - Mmcorc /Id# 202099, Saint Louis Park, Minnesota
  - Washington University School /ID# 200621, St Louis, Missouri
  - University of Nebraska /ID# 203195, Omaha, Nebraska
  - The Valley Hospital /ID# 169999, Paramus, New Jersey
  - Duke University Medical Center /ID# 169657, Durham, North Carolina
  - Fairview Hospital - Moll Pavilion /ID# 205910, Cleveland, Ohio
  - Cleveland Clinic Main Campus /ID# 200325, Cleveland, Ohio
  - Hillcrest Hospital /ID# 205911, Mayfield Heights, Ohio
  - INTEGRIS Cancer Institute of OK/INTEGRIS Southwest Medical Center /ID# 200831, Oklahoma City, Oklahoma
  - INTEGRIS Cancer Institute /ID# 200832, Oklahoma City, Oklahoma
  - Oregon Health and Science University /ID# 170807, Portland, Oregon
  - Thomas Jefferson University /ID# 200833, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Ctr /ID# 200672, Pittsburgh, Pennsylvania
  - Greenville Hospital System /ID# 203021, Greenville, South Carolina
  - Tennessee Oncology-Nashville Centennial /ID# 203424, Nashville, Tennessee
  - Tennessee Oncology, PLLC /ID# 203581, Nashville, Tennessee
  - Ut Southwestern Medical Center /Parkland Health and Hospital System /Id# 210112, Dallas, Texas
  - UTSW-Dallas /ID# 204031, Dallas, Texas
  - Millennium Oncology /ID# 204925, Houston, Texas
  - Virginia Cancer Specialists /ID# 169293, Fairfax, Virginia
  - Kadlec Clinic Hematology and O /ID# 170811, Kennewick, Washington
  - Medical Oncology Associates /ID# 169290, Spokane, Washington
  - Univ of Wisconsin Hosp/Clinics /ID# 200424, Madison, Wisconsin
- Belgium (5):
  - UZ Gent /ID# 200691, Ghent, Oost-Vlaanderen
  - Imelda Ziekenhuis /ID# 200693, Bonheiden
  - Cliniques universitaires Saint /ID# 203101, Brussels
  - UZ Antwerp /ID# 200694, Edegem
  - UZ Leuven /ID# 200001, Leuven
- Canada (2):
  - Hospital Maisonneuve-Rosemont /ID# 171590, Montreal, Quebec
  - Jewish General Hospital /ID# 171584, Montreal, Quebec
- South Korea (4):
  - National Cancer Center /ID# 170879, Goyang, Gyeonggido
  - Samsung Medical Center /ID# 170875, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 170878, Seoul
  - Asan Medical Center /ID# 170877, Seoul
- Spain (5):
  - Hospital Universitario Vall d'Hebron /ID# 200186, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 200189, Madrid
  - Hospital Clinico Universitario San Carlos /ID# 201721, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 200187, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 200190, Madrid
- Taiwan (3):
  - National Taiwan Univ Hosp /ID# 170677, Taipei City, Taipei
  - Taichung Veterans General Hosp /ID# 170123, Taichung
  - Taipei Veterans General Hosp /ID# 170675, Taipei

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Strickler JH, Cubillo A, Liang JT, Matrana M, Kozloff M, Lowe T, Blaney M, Sahtout M, Naumovski L, Wainberg ZA. Efficacy and safety of dilpacimab (ABT-165) versus bevacizumab plus FOLFIRI in metastatic colorectal cancer: a phase II study. Future Oncol. 2022 Sep;18(27):3011-3020. doi: 10.2217/fon-2021-1603. Epub 2022 Aug 3. PMID 35920133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The intent to treat (ITT) population included all randomized participants and was used for all efficacy and baseline analyses.
Pre-assignment Details: A total of 70 participants were randomized to 1 of the 2 study treatments. Participants were grouped according to treatment as randomized.
Groups:
- ABT-165 Plus FOLFIRI: ABT-165 plus FOLFIRI (irinotecan, leucovorin, fluorouracil) IV infusion for a 14 day cycle until disease progression or intolerable toxicity
- Bevacizumab Plus FOLFIRI: Bevacizumab plus FOLFIRI (irinotecan, leucovorin, fluorouracil) IV infusion for a 14 day cycle until disease progression or intolerable toxicity
Period: Overall Study
Arm/Group | ABT-165 Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Started | 36 | 34
Completed | 0 | 0
Not Completed | 36 | 34
Not completed — Withdrew Consent | 5 | 4
Not completed — Death | 12 | 6
Not completed — Study terminated by Sponsor | 18 | 23
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-165 Plus FOLFIRI | Bevacizumab Plus FOLFIRI | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (11.41) | 60.2 (10.19) | 60.5 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 21 | 19 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 34 | 31 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 20 | 40
  Black or African American | 2 | 1 | 3
  Asian | 11 | 11 | 22
  American Indian or Alaska native | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Missing | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization until the first occurrence of radiographic progression determined by investigator assessment or death from any cause.
Time Frame: Follow up continued until the first occurrence of radiographic progression, death from any cause or termination of the study; median follow-up time was 25.6(0.3-64.4) and 37.6(0.3-66.3) weeks in ABT-165 plus FOLFIRI and Bevacizumab + FOLFIRI, respectively
Population: Intent to Treat (ITT): includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ABT-165 Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Number analyzed (Participants) | 36 | 34
Months | 3.78 [2.07 to 7.20] | 7.36 [5.68 to 10.55]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the proportion of participants with a complete response (CR) or partial response (PR) as determined by a investigator assessment based on Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1.
Time Frame: From randomization up to 30 days after last dose of study drug; median time on follow-up was 25.6 (0.3 - 64.4) and 37.6 (0.3 - 66.3) weeks in ABT-165 plus FOLFIRI and Bevacizumab plus FOLFIRI, respectively
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-165 Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Number analyzed (Participants) | 36 | 34
percentage of participants | 5.6 [0.7 to 18.7] | 14.7 [5.0 to 31.1]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization until death from any cause.
Time Frame: as for outcome 1
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ABT-165 Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Number analyzed (Participants) | 36 | 34
Months | 7.95 [7.00 to NA] — Due to early termination of the study, there was insufficient follow-up time, which limited estimates of OS. | NA [10.55 to NA] — Due to early termination of the study, there was insufficient follow-up time, which limited estimates of OS.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study drug to 90 days (+15 days) after the last dose and then every 90 days (+15 days) throughout the survival period;the median duration across both treatment groups was 38.6 (3.0-99.3) weeks.
Arm/Group | ABT-165 Plus FOLFIRI | Bevacizumab Plus FOLFIRI
All-Cause Mortality (participants affected / at risk) | 12/34 | 6/32
Serious Adverse Events (participants affected / at risk) | 17/34 | 8/32
Other Adverse Events (participants affected / at risk) | 32/34 | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-165 Plus FOLFIRI (N=34) | Bevacizumab Plus FOLFIRI (N=32)
ANAEMIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 2 (2) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
DISEASE PROGRESSION (General disorders) | 0 (0) | 1 (1)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
ANAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
HEPATITIS B (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 2 (2) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-165 Plus FOLFIRI (N=34) | Bevacizumab Plus FOLFIRI (N=32)
ANAEMIA (Blood and lymphatic system disorders) | 3 (4) | 5 (10)
LEUKOPENIA (Blood and lymphatic system disorders) | 5 (12) | 5 (7)
NEUTROPENIA (Blood and lymphatic system disorders) | 14 (31) | 12 (32)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (5) | 2 (2)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 2 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 6 (7) | 6 (7)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 4 (5)
ANAL FISSURE (Gastrointestinal disorders) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 8 (8) | 5 (10)
DIARRHOEA (Gastrointestinal disorders) | 18 (23) | 15 (20)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 3 (3)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 4 (4)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 3 (3)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 18 (25) | 14 (19)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (3)
STOMATITIS (Gastrointestinal disorders) | 7 (7) | 10 (14)
TOOTH LOSS (Gastrointestinal disorders) | 2 (2) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 2 (2)
VOMITING (Gastrointestinal disorders) | 5 (12) | 9 (14)
ASTHENIA (General disorders) | 2 (2) | 2 (2)
CATHETER SITE PAIN (General disorders) | 2 (2) | 0 (0)
CHILLS (General disorders) | 2 (2) | 0 (0)
FATIGUE (General disorders) | 14 (18) | 13 (24)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 2 (8)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 4 (4) | 0 (0)
PYREXIA (General disorders) | 3 (3) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 3 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 5 (5)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 4 (4)
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 (0) | 2 (2)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (1) | 3 (4)
NEUTROPHIL COUNT DECREASED (Investigations) | 4 (8) | 2 (5)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 3 (4)
WEIGHT DECREASED (Investigations) | 1 (1) | 3 (3)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2 (2) | 2 (2)
DECREASED APPETITE (Metabolism and nutrition disorders) | 8 (8) | 7 (9)
DEHYDRATION (Metabolism and nutrition disorders) | 6 (6) | 3 (4)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 5 (5) | 2 (3)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2)
DIZZINESS (Nervous system disorders) | 7 (8) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 3 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 6 (6) | 4 (4)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 3 (3)
ANXIETY (Psychiatric disorders) | 4 (4) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 4 (4)
INSOMNIA (Psychiatric disorders) | 0 (0) | 4 (4)
PROTEINURIA (Renal and urinary disorders) | 2 (2) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 2 (2) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
HYPERTENSION (Vascular disorders) | 10 (15) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT03368859/Prot_SAP_000.pdf